CLINICAL TRIAL: NCT04461197
Title: Efficacy of the Therapeutic Effects of Adjunctive Treatment of Plantar Orthoses With Extracorporeal Shock Wave Therapy in Plantar Fasciitis: a Randomized Clinical Trial.
Brief Title: Efficacy of the Treatment of Plantar Orthoses With Extracorporeal Shock Wave Therapy in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, MANUEL PABON CARRASCO, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRESEUE-Foot 2
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Fasciitis, Plantar, Chronic
Keywords: Fasciitis, Plantar; Foot Orthoses; High-Energy Shock Waves
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT + orthotic insole (Experimental): (shock waves + orthotic insole +Stretches of the posterior muscle chain)
  Interventions: Device: customised foot orthoses
- ESWT + flat insole (Placebo Comparator): (shock waves + flat insole + Stretches of the posterior muscle chain)
  Interventions: Device: orthotic insole

INTERVENTIONS:
Device: customised foot orthoses — The foot orthoses for group A were custom made using phenolic foam molds of the feet. Separated molds were made of both feet for all the participants. . The insole was made based on a positive mold of plaster with 45 Shore cork materials with horizontal thrusts just proximal to the metatarsal heads, with the intention of correcting the pathological subtalar pronation, with a 3mm bilateral raising of the heel and a bilateral latex metatarsal bar.
  Arms: ESWT + orthotic insole
Device: orthotic insole — For group B, a flat insole of polyester resin was made, fitting it to the foot's size.
  Arms: ESWT + flat insole

SUMMARY:
Plantar fasciitis is inflammation of plantar fascia. It arises from degeneration and chronic inflammation. Treatment of plantar fasciitis contains conservative methods like rest, body weight control, stretching exercise, non-steroidal anti-inflammatory drugs and arch supports. ESWT has commonly been used for the treatment of plantar fasciitis. The shock waves can be radial or focused. The aim of this study was to evaluate the effectiveness of the adjuvant use of plantar orthoses in the process of plantar fasciitis when extracorporeal shock waves are applied. The hypothesis porposed was that the use of extracorporeal shock waves together with the use of custom foot orthotics improves the symptoms produced by plantar fasciitis. This study is planned as double-blind, randomized controlled trial. Participants are randomly allocated to two groups: the ESWT group and the custom foot orthotics and ESWT group. Radial ESWT will be applied in this study.

The people receiving the therapy and the people assessing the outcomes are blinded . Both group will recieve ESWT one session per week for three weeks. Each session will last for 2-5 minutes. The primary outcome measure of this study is change in heel pain of affected side assessed using Visual Analog Scale. The secondary outcome measure is Roles y Maudsley scores. The primary endpoint of this study is to determine a decrease in pain score according to Visual Analog Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 65 years
* able to understand the explanations about the potential benefits and risks of participating in the study
* both genders
* diagnosis of chronic plantar fasciitis
* duration of symptoms equal or superior to 6 months at the time of enrollment
* Foot Posture Index ≥ +6 (pronated foot in one or both feet).

Exclusion Criteria:

* being younger than 18 years of age
* previous treatments with shock wave devices
* previous surgery on the painful heel; history of calcaneus fracture
* any inflammation at the level of the ankle
* infection in the treated area
* patients with diabetes mellitus or cardiac or respiratory disease
* osteomyelitis
* patients on anticoagulant drugs
* pregnancy
* patients on immunosuppressive therapy
* rheumatoid arthritis or history of rheumatic disease
* neurological deficits
* malignant disease with or without metastases
* significant liver function abnormalities
* neurological or vascular insufficiency in the painful heel; fasciotomy or heel spur surgery
* discrepancy in the length of the foot > 5 mm; previous back of foot surgery
* patients treated with rigid plantar supports

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | Baseline
  Heel pain intensity was referred to as 0-10, in which 0= no pain at all and 10= the worst pain possible

SECONDARY OUTCOMES:
Roles-Maudsley (RM) scores | Baseline
  This is a self-administered scale of functional valuation which classifies the patients into 4 categories

CONTACTS AND LOCATIONS:
Overall Officials: Ana J Perez, Dra., Study Director — University of Seville
Locations (1):
- Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No